CLINICAL TRIAL: NCT04350840
Title: Performance of Real-time Optical Diagnosis for Colon Polyp According to the Confidence Rate of Endoscopists
Brief Title: Seoul National University Hospital Gangnam-Real Time Optical Diagnosis Program 2: Gangnam-READI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: H-2001083-1095
Record Dates: First submitted 2020-03-22; First posted 2020-04-17 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feedback (Experimental): Participating endoscopists will make high confidence diagnosis according to their judgment time
  Interventions: Behavioral: feedback

INTERVENTIONS:
Behavioral: feedback — feedback of optical diagnosis performance per 3 month

SUMMARY:
Accurate optical diagnosis of colorectal polyps could allow a "resect and discard" strategy based on the results of the optical biopsy. Even though intensive training for optical diagnosis, there is still wide variability in individual endoscopists to meet the PIVI thresholds. The investigators with experience of prior optical diagnosis training perform new education and drill to apply proper high confidence according to their decision time. After the education program, the investigators prospectively evaluate real-time optical biopsy analysis of polyps in 8 academic gastroenterologists.

DETAILED DESCRIPTION:
This study is an extension of the Gangnam-READI program (NCT02516748) in Seoul National University Hospital Healthcare System Gangnam Center. This study is composed of two periods. First, an education program on predicting polyp histology and real-time optical diagnosis will be performed by 8 endoscopists From February to March 2020. In the second period from April 2020 till October 2020(total 6 months), real-time optical diagnosis with time drill for diminutive and small colorectal polyps will be activated. Endoscopists will have 3 seconds rule to make high confidence diagnosis and have feedbacks on their accuracy of optical diagnosis for polyps per 3 months. The performance will be evaluated by comparing the optically predicted diagnosis with the actual histologic diagnosis. Negative predictive value for the prediction of non-neoplastic polyp and concordance of surveillance intervals for diminutive polyps diagnosed optically with high confidence will be measured. In addition, the characteristics of the endoscopist affecting the performance of optical diagnosis were investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified gastroenterologists
2. Endoscopists who finished ex-vivo optical diagnosis training

Exclusion Criteria:

1. Inflammatory bowel disease
2. Previous colon cancer history
3. Previous colon op. history
4. Melanosis coli

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
PIVI threshold | 12 months
  Negative predictive value for the prediction of nonneoplastic polyp and concordance of surveillance intervals for diminutive polyps diagnosed optically with high confidence

CONTACTS AND LOCATIONS:
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae JH, Lee C, Kang HY, Kwak MS, Doo EY, Seo JY, Song JH, Yang SY, Yang JI, Lim SH, Yim JY, Lim JH, Chung GE, Chung SJ, Jin EH, Park B, Kim JS. Improved Real-Time Optical Diagnosis of Colorectal Polyps Following a Comprehensive Training Program. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2479-2488.e4. doi: 10.1016/j.cgh.2019.02.019. Epub 2019 Feb 14. PMID 30772588
- [Derived] Kim J, Lim SH, Kang HY, Song JH, Yang SY, Chung GE, Jin EH, Choi JM, Bae JH. Impact of 3-second rule for high confidence assignment on the performance of endoscopists for the real-time optical diagnosis of colorectal polyps. Endoscopy. 2023 Oct;55(10):945-951. doi: 10.1055/a-2073-3411. Epub 2023 May 12. PMID 37172938